CLINICAL TRIAL: NCT07117162
Title: Increasing Access to Care: An Advanced Virtual Care Delivery Protocol to Deliver Diagnostic and Therapeutic Services to Underserved Veterans With ADRD
Brief Title: Improving Access to Care for Veterans With Memory Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1850695
Record Dates: First submitted 2025-07-25; First posted 2025-08-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADRD Care Delivery Protocol (Experimental): Patients will undergo telehealth preparedness assessment, cognitive screening, and blood biomarker testing prior to the initial consultation with the specialist.
  Interventions: Other: ADRD Care Delivery Protocol
- Usual Care (No Intervention): Patients will undergo usual care with all evaluation and testing at the discretion of the specialist.

INTERVENTIONS:
Other: ADRD Care Delivery Protocol — 1. Included in arm/group descriptions
  Arms: ADRD Care Delivery Protocol

SUMMARY:
This study evaluates a care delivery protocol to improve access to care for Veterans with Alzheimer's Disease and Related Disorders (ADRD). A randomized controlled trial will enroll Veterans with mild cognitive impairment or early dementia at VA Pittsburgh. The ADRD care delivery protocol integrates telehealth, advanced diagnostics, and streamlined workflows to expedite screening for eligibility for amyloid targeting therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild cognitive impairment or mild dementia due to suspected or confirmed AD with a 5 minute telephone MoCA score >7
* Meets VA MUE inclusion/exclusion criteria for mAb therapy for AD
* Enrolled in VA care
* Lives in a home setting (i.e., not in an institutional setting such as a nursing home, Community Living Center, or hospital)
* Has a working telephone
* 18 years and older
* Able to communicate in English
* Willing to give informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time to Eligibility Determination | From date of randomization until the date of determination of eligibility for monoclonal antibody therapy, assessed up to 12 months.
  Compare the number of days from randomization to the determination of eligibility for monoclonal antibody therapy for both the intervention and usual care groups, assessed up to 12 months.
Time to Initial Infusion | From date of randomization until the date of first infusion, assessed up to 12 months.
  Compare the number of days from the date of randomization to the initial infusion of monoclonal antibody therapy for both the intervention and usual care groups, assessed up to 12 months.

SECONDARY OUTCOMES:
Number of Participants and Instances of Additional testing | 1 year
  Chart review will be used to determine the number of participants who underwent additional testing and the total number of additional tests performed. This includes counting instances of APOE genetic testing, MRI brain imaging, and amyloid PET imaging as ordered at the discretion of the specialist.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DONANEMAB-AZBT INJ,SOLN - VA Formulary Advisor. Accessed December 12, 2024. https://www.va.gov/formularyadvisor/drugs/4043274-DONANEMAB-AZBT-INJ-SOLN
- [Background] LECANEMAB-IRMB INJ,SOLN - VA Formulary Advisor. Accessed December 12, 2024. https://www.va.gov/formularyadvisor/drugs/4041980-LECANEMAB-IRMB-INJ-SOLN
- [Background] Sims JR, Zimmer JA, Evans CD, Lu M, Ardayfio P, Sparks J, Wessels AM, Shcherbinin S, Wang H, Monkul Nery ES, Collins EC, Solomon P, Salloway S, Apostolova LG, Hansson O, Ritchie C, Brooks DA, Mintun M, Skovronsky DM; TRAILBLAZER-ALZ 2 Investigators. Donanemab in Early Symptomatic Alzheimer Disease: The TRAILBLAZER-ALZ 2 Randomized Clinical Trial. JAMA. 2023 Aug 8;330(6):512-527. doi: 10.1001/jama.2023.13239. PMID 37459141
- [Background] Mintun MA, Lo AC, Duggan Evans C, Wessels AM, Ardayfio PA, Andersen SW, Shcherbinin S, Sparks J, Sims JR, Brys M, Apostolova LG, Salloway SP, Skovronsky DM. Donanemab in Early Alzheimer's Disease. N Engl J Med. 2021 May 6;384(18):1691-1704. doi: 10.1056/NEJMoa2100708. Epub 2021 Mar 13. PMID 33720637
- [Background] Yaffe K, Vittinghoff E, Lindquist K, Barnes D, Covinsky KE, Neylan T, Kluse M, Marmar C. Posttraumatic stress disorder and risk of dementia among US veterans. Arch Gen Psychiatry. 2010 Jun;67(6):608-13. doi: 10.1001/archgenpsychiatry.2010.61. PMID 20530010
- [Background] Walker LE, Poltavskiy E, Janak JC, Beyer CA, Stewart IJ, Howard JT. US Military Service and Racial/Ethnic Differences in Cardiovascular Disease: An Analysis of the 2011-2016 Behavioral Risk Factor Surveillance System. Ethn Dis. 2019 Jul 18;29(3):451-462. doi: 10.18865/ed.29.3.451. eCollection 2019 Summer. PMID 31367165
- [Background] 2024 Alzheimer's disease facts and figures. Alzheimers Dement. 2024 May;20(5):3708-3821. doi: 10.1002/alz.13809. Epub 2024 Apr 30. PMID 38689398
- [Background] VHA_ALZHEIMERS_DEMENTIA_Statistical_Projections_FY21_and_FY33_sgc121820.pdf. Accessed December 12, 2024. https://www.va.gov/GERIATRICS/docs/VHA_ALZHEIMERS_DEMENTIA_Statistical_Projections_FY21_and_FY33_sgc121820.pdf
- [Background] Swanson CJ, Zhang Y, Dhadda S, Wang J, Kaplow J, Lai RYK, Lannfelt L, Bradley H, Rabe M, Koyama A, Reyderman L, Berry DA, Berry S, Gordon R, Kramer LD, Cummings JL. A randomized, double-blind, phase 2b proof-of-concept clinical trial in early Alzheimer's disease with lecanemab, an anti-Abeta protofibril antibody. Alzheimers Res Ther. 2021 Apr 17;13(1):80. doi: 10.1186/s13195-021-00813-8. PMID 33865446